CLINICAL TRIAL: NCT07144904
Title: A Side-Randomized, Self-Controlled Trial Assessing the Efficacy of Indocyanine Green Fluorescence Imaging for Intraoperative Ureter Identification During Robot-Assisted Single-Site Surgery in Advanced-Stage Endometriosis
Brief Title: Assessing the Efficacy of Indocyanine Green for Ureter Identification During Robot-Assisted Surgery in Advanced-Stage Endometriosis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, XIAOMING GUAN, Division Chief of Minimally Invasive Gynecologic Surgery, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: H-57801
Record Dates: First submitted 2025-08-14; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Indocyanine Green (ICG); Robotic Surgical Procedure; Deep Infiltrating Endometriosis (DIE); Endometriosis Pelvic; Endometriosis (Diagnosis); Endometriosis of the Cul-de-sac; Ureteral Stent Placement; Ureteral Injury; Endometriosis Ovaries
Keywords: ureteral stent placement; indocyanine green; endometriosis; robotic surgery; ureteral identification
MeSH Terms: conditions — Endometriosis; Disease | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: This study will be a side-randomized, self-controlled trial where participant will be randomized to receive ICG-assisted ureteral identification on either the left or right side. Randomization will be conducted using a computer-generated block randomization method. No stratification based on preoperative characteristics is planned.The patient will be blinded to their randomization, and the surgeon will be initially blinded as well. Ureteral ICG stent placement will be performed after anesthesia induction and while the surgeon is scrubbing. The assistant surgeon, surgical staff, research assistants, and statisticians will not be blinded.
Who Masked: Participant
Masking Description: Participants will be informed that the study involves intraoperative indocyanine green (ICG)-assisted ureter identification and that they will be randomized to receive a temporary ICG ureteral stent on either the left or right side. They will be advised that there is a 50% probability of assignment to either side and that they will remain blinded to their allocation throughout the study. Risks and potential benefits of the procedure will be explained, and written informed consent will be obtained. Each participant will be assigned a unique study number for data de-identification prior to randomization, which will be conducted using a computer-generated sequence in REDCap. The operating surgeon will be informed of the assigned side.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: ICG-Assisted Ureteral Identification (Unilateral) (Experimental): Participants assigned to this study will undergo intraoperative ureteral identification using indocyanine green (ICG) fluorescence imaging in either left or right side. A temporary ureteral stent will be inserted on the randomized side (left or right) prior to ureterolysis and endometriosis resection. ICG will be administered through the stent to facilitate real-time fluorescence visualization of the ureter during robot-assisted single-site surgery. The contralateral side will serve as the control arm (standard visualization without ICG).
  Interventions: Drug: Indocyanine Green (ICG)-Assisted Ureteral Identification
- Arm B: Standard Visualization (Contralateral Control) (Active Comparator): Participants assigned to this study will undergo intraoperative ureteral identification using indocyanine green (ICG) fluorescence imaging in either left or right side. A temporary ureteral stent will be inserted on the randomized side (left or right) prior to ureterolysis and endometriosis resection. ICG will be administered through the stent to facilitate real-time fluorescence visualization of the ureter during robot-assisted single-site surgery. The contralateral side will serve as the control arm (standard visualization without ICG).
  Interventions: Procedure: Standard Ureteral Identification without ICG

INTERVENTIONS:
Drug: Indocyanine Green (ICG)-Assisted Ureteral Identification — A temporary ureteral stent will be placed unilaterally (left or right) prior to robotic procedures in participants undergoing robot-assisted single-site surgery for advanced-stage endometriosis. Indocyanine green (ICG) will be administered through the stent to enable real-time fluorescence imaging for intraoperative ureter identification. The contralateral ureter will be identified using standard visualization techniques without ICG. Side allocation (ICG vs. control) will be determined by computer-generated block randomization.
  Arms: Arm A: ICG-Assisted Ureteral Identification (Unilateral)
Procedure: Standard Ureteral Identification without ICG — Ureter identification will be performed using standard intraoperative visualization techniques without the use of indocyanine green (ICG) fluorescence imaging. This will be done on the contralateral side to the randomized ICG-assisted ureteral identification during robot-assisted single-site surgery for advanced-stage endometriosis.
  Arms: Arm B: Standard Visualization (Contralateral Control)

SUMMARY:
The goal of this side-randomized, self-controlled trial, 1-site study is to explore the efficacy of Indocyanine Green Fluorescence (ICG) for Intraoperative Ureter Identification During Robot-Assisted Single-Site Surgery in Advanced-Stage Endometriosis.

Researchers will perform temporary ureteral stent using indocyanine green fluorescence for intraoperative ureteral identification on either the left or right side of subjects who are undergoing a robotic assisted transumbilical resection of advanced endometriosis.

Participants will be randomized to receive ICG-assisted ureteral identification on either the left or right side. Randomization will be conducted using a computer-generated block randomization method.

The primary aim is to determine whether ICG-assisted ureter visualization can reduce operative time for endometriosis resection and ureterolysis, and minimize the risk of ureteral injury.

Secondary objectives are to assess the feasibility and safety of temporary ureteral ICG stenting for intraoperative ureter identification in advanced endometriosis.

DETAILED DESCRIPTION:
Clinic schedules will be screened for possible surgical candidates by the attending surgeons, fellow, and research assistant. Patients will be recruited from the minimally invasive gynecologic surgery clinics of Dr. Guan. Patients who are meet the inclusion and exclusion criteria will undergo recruitment and be offered to participate in the research study. The research study will be introduced by the surgeon (Dr. Guan) during their pre-operative consultation. If the patient is interested in hearing more about the study and possibly participating, then the investigators will interact with the patient in order to explain the study in detail, answer questions, and obtain informed consent. Patients will be able to learn more about the study and provide consent in-person (after their initial surgical consultation is completed but prior to leaving clinic), through remote consent via telephone, or on the day of surgery. This should allow the patient sufficient time to evaluate the risks and benefits of participation and ensure informed consent or informed refusal of participation, minimizing coercion. Participants will be counseled that their consent or refusal to participate will not otherwise alter their routine perioperative care or surgery.

After the patient was prepped and draped, a 17F sheathed cystoscope was threaded with a single 5F open-ended 27 cm stent. Twenty-five mg of ICG was diluted with 10 ml of normal saline and placed on the lur-lock of a single open-ended stent. The cystoscope was primed. Time was started once the labia were parted to find the urethra. The cystoscope was advanced into the bladder, and both ureteral openings were visualized before placement of the singular stent. The side randomized by computer to receive ICG was again visualized, and the stent was advanced retrograde to a depth of 15 cm. Five ml of ICG was then injected into the stent. The stent was allowed to sit in the same ureter for 60 seconds before the stent and cystoscope were removed. Once all instruments were removed from the urethra, time was stopped and recorded.

Once the robot was docked, the camera was positioned to visualize both pelvic sidewalls. At this point, the surgeon remained blinded to the side injected with ICG. Ureter identification was then performed by the both the surgeon and fellows on each side, and the time required to identify each ureter was recorded. After identification, they rated the difficulty of ureteral dissection on each side using a visual analog scale (VAS), where 0 indicated extremely easy and 10 indicated maximal difficulty, based on anatomical complexity and the extent of adhesions.

When the surgeon begins pelvic sidewall endometriosis resection, timing will be initiated to record the duration of each step and the total operative time for each side. The side without ICG injection will be addressed first. The procedures will follow a standardized sequence: lysis of adhesions - ureterolysis -endometriosis resection.

Following the surgery, the surgeon is required to complete the Surgery Task Load Index (SURG-TLX) for each side.

Data regarding the participant's demographics and pre-operative symptoms will be collected through standardized questionnaires administered in clinic that have been validated for use in endometriosis participants. It will also be collected from routine pre-operative data that is standardly recorded in clinical documentation and will be extracted from the electronic medical record (EPIC).

Intra-operative data will be extracted from the electronic medical record (EPIC) or recorded during the OR case by the operating room circulator nurse or research assistant. Post-operative data will be collected from the electronic medical record.

Sample Size：Using a paired t-test or Wilcoxon signed-rank test presuming d = 0.5 (a medium Cohen's d effect size), α = 0.05, power = 0.80, and self-control, the total sample size required is 35. Accounting for a 10% dropout, that would be 39 per group. Thus, the investigators will recruit until the investigators have achieved 40 participants per group.

Statistical Analysis: 1. Descriptive statistics were generated. Continuous variables were tested for normality with the Kolmogorov-Smirnov test. Normal distribution variables are shown as mean±standard deviation (SD), with non-normal distribution data described as median [inter-quartile range (IQR)]. Categorical data are reported as proportions and percentages. 2. Total operative time of each side, and operative time of every procedures, ureter identification time without ICG and VAS score will be compared between two sides using the paired t-test or paired Wilcoxon signed rank test as appropriate. 3. All statistical analysis was carried out using SPSS version 25 (Inc, Chicago, IL, USA). Statistical significance was set at P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Stage III or IV endometriosis (rASRM classification)
* Planned robotic transabdominal endometriosis excision with or without hysterectomy.

Exclusion Criteria:

- Subjects who are part of a vulnerable population will be excluded including those who are prisoners, younger than 18 years old, pregnant, individuals with mental disabilities or cognitive impairment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Comparison of operative time between the ICG-assisted and standard visualization sides | Intraoperative, measured during the surgical procedure on the day of surgery.
  Total operative time was calculated for each side, as well as for each individual procedure. The total operative time represents the sum of the operative times for all individual procedures performed.

SECONDARY OUTCOMES:
Incidence of ureter or bladder symptoms or complications & Surgical complication rate by Clavien-Dindo classification | Postoperative, up to 6 weeks after surgery.
  Number and percentage of participants with postoperative ureter or bladder-related symptoms or complications, confirmed by clinical evaluation.Number and percentage of participants experiencing surgical complications, graded according to the Clavien-Dindo classification system.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Guan, PhD, MD, Principal Investigator — Department Chair of Minimally Invasive Gynecologic Surgery
Locations (1):
- Texas Childrens Hospital Pavilion for Women, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No